CLINICAL TRIAL: NCT06112132
Title: National Observatory of Children Hospitalized for Bronchiolitis
Acronym: OVNI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Association Clinique Thérapeutique Infantile du val de Marne (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: OVNI
Record Dates: First submitted 2023-10-27; First posted 2023-11-01 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2023-10

CONDITIONS: Bronchiolitis
MeSH Terms: conditions — Bronchiolitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is an observational, multicenter and prospective study for surveillance of case of hospitalised children for bronchiolitis associated or not to RSV or other viruses (isolated or associated with RSV)

DETAILED DESCRIPTION:
The aim of this surveillance is to observe and describe the cases hospitalized for bronchiolitis in the 2023/2024 season in the context of routine immunization with Nirsevimab.

ELIGIBILITY:
Inclusion Criteria:

* Children under 12 months of age
* In one of the 6 study sites
* From October 15, 2023
* For acute bronchiolitis defined according to current national and international recommendations
* Hospitalized from the pediatric emergency department.

Exclusion Criteria:

- Refusal to participate by patient relative or legal representative

Ages: 1 Day to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children hospilalized for bronchiolitis
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2023-10-15 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of patients hospitalized for bronchiolitis | 1 year
  Assessment of the number of hospitalized bronchiolitis in the context of routine immunization with Nirsevimab

SECONDARY OUTCOMES:
Proportion of RSV vs non-RSV associated to bronchiolitis hospitalizations | 1 year
  Assessment of proportion of RSV vs non- RSV associated bronchiolitis hospitalizations
Proportion of other viruses associated to bronchiolitis hospitalizations. | 1 year
  Assessment of the proportion of other viruses (isolated or associated with RSV) associated bronchiolitis hospitalizations
Proportion of patients immunized with Nirsevimab among children hospitalized for bronchiolitis | 1 year
  Description of immunization status with Nirsevimab of hospitalized patients for bronchiolitis overall (RSV+, RSV-) and other viruses (isolated or associated with RSV)
Proportion of demographics and clinical characteristics of patients hospitalized for bronchiolitis overall | 1 year
  Description of demographics (including immunization status with Nirsevimab) and clinical characteristics of patients hospitalized for bronchiolitis overall ( RSV+, RSV-) and other viruses (isolated or associated with RSV)
Proportion of demographics, clinical and viral characteristics of patients hospitalized for bronchiolitis requiring ventilation support | 1 year
  Description of demographics (including immunization status with Nirsevimab), clinical and viral characteristics of patients hospitalized for bronchiolitis requiring ventilation support
Length of hospital stay of children with bronchiolitis overall in France | 1 year
  Assesment of the duration of hospitalization for bronchiolitis overall (RSV+, RSV-) in France
Length of hospital stay of children with bronchiolitis in France according to immunization status with Nirsevimab | 1 year
  Assesment of the duration of hospitalization for bronchiolitis according to immunization status with Nirsevimab

CONTACTS AND LOCATIONS:
Overall Officials: Levy Corinne, Study Director — Association Clinique Thérapeutique Infantile du val de Marne; Jeziorski Eric, Principal Investigator — CHU Montpellier, Service Urgence et Post-urgences pédiatrique
Locations (1):
- ACTIV, Créteil, France

REFERENCES:
- [Derived] Jeziorski E, Ouziel A, Cotillon M, Bridonneau C, Bizot E, Basse C, Portefaix A, Dubos F, Bechet S, Domitien L, Jaillet C, Abrudan S, Kramer R, Gajdos V, Launay E, Basmaci R, Gillet Y, Cohen R, Levy C. Impact of Nirsevimab on Respiratory Syncytial Virus Bronchiolitis in Hospitalized Infants: A Real-World Study. Pediatr Infect Dis J. 2025 Apr 1;44(4):e124-e126. doi: 10.1097/INF.0000000000004630. Epub 2024 Nov 26. PMID 39589139